CLINICAL TRIAL: NCT05530174
Title: The Effect of Single vs Multiple Prophylactic Antibiotic Doses on PJI Following Primary THA in Patients With a Fracture: A Cross-over, Cluster Randomized Controlled, Non-inferiority Trial Based on National Quality Databases: ProHipQ-F
Brief Title: Effect of Single vs Multiple Prophylactic Antibiotic Doses on PJI Following Primary THA in Patients With a Fracture
Acronym: ProHipQ-F
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soren Overgaard (Other)
Collaborators: University of Copenhagen (Other); University Hospital Bispebjerg and Frederiksberg (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); University of Aarhus (Other); Sygehus Lillebaelt (Other)
Responsible Party: Sponsor-Investigator, Soren Overgaard, Clinical Professor, DMSc, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ProHipQ Fracture
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Fracture of Hip; Total Hip Arthroplasty; Prosthetic-joint Infection; Fracture Acetabular
Keywords: Antibiotic Prophylaxis; Hip Fracture; Acetabular Fracture; Total Hip Replacement; Total Hip Arthroplasty; Prosthetic Joint Infection; PJI; Cluster Randomized Controlled Trial; Randomized Controlled Trial; RCT; THA
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: The Pro-Hip-Quality Trial is a Cluster Randomized Trial with an embedded Cross-Over Design where each clinical center (C: 1, 2, 3, …., 36 individual sites) will be running a specific intervention (i.e. single- or multiple-dose antibiotics) throughout 12 months, and the subsequent year the clinical department will automatically switch to the opposite intervention (i.e. multiple- or single-dose antibiotics).
Masking Description: Blinding will not be applicable, because it is considered infeasible to expose participants and clinical personnel to this in either of the groups since any specific clinic will follow their allocated specific (single- or multiple-dose) routine during an entire 1-year period and their routine treatment of any complication (before switching).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A, Single-dose practice (Experimental): One preoperative single dose of either Dicloxacillin/Cloxacillin 2g OR Cefuroxime 1.5g administered intravenously prior to surgical incision.
  As the study is a non-inferiority trial, we have chosen the Experimental design category.
  Interventions: Other: Antibiotic dosage practice
- Treatment B, Multiple-dose practice (Active Comparator): One preoperative dose of either Dicloxacillin/Cloxacillin 2g OR Cefuroxime 1.5g administered intravenously prior to surgical incision followed by 3 postoperative doses of Dicloxacillin/Cloxacillin 1g x 3 OR Cefuroxime 750mg x 3 within 24 hours after the preoperative dose.
  Interventions: Other: Antibiotic dosage practice

INTERVENTIONS:
Other: Antibiotic dosage practice — Patient inclusion starts day one, cross-over of departments from treatment A (single-dose) to B (multiple-dose) or vice versa after one year and end of inclusion happens after 2 years.
  All centers in Denmark use either Cloxacillin/Dicloxacillin, Cefuroxime or both drugs as standard prophylactic antibiotic practice for THA. In cases of cephalosporin allergy or general beta lactam allergy, the antibiotic clindamycin may be administered.
  In this trial, patients will be administered the standard prophylactic antibiotic practice of either single-dose (A) or multiple-doses (B) of antibiotics administered at each respective cluster that respective year. Both practices of dose administration for antibiotic prophylaxis (i.e. single- or multiple-dose) follow current standards of treatment and are based on present clinical practice guidelines.

SUMMARY:
Aim: To compare the effect of one single dose versus multiple doses of prophylactic antibiotics administered within 24 hours, on the development of PJI after surgery in patients undergoing primary THA due to an acute fracture or sequelae of proximal femoral or acetabular fractures.

The study is designed as a cross-over, cluster randomized, non-inferiority trial. All Danish orthopedic surgery departments performing primary THA with the majority being within inclusion criteria will be involved: Based on national quality databases, two-year cohorts of approximately 2,000 primary THAs due to a fracture or sequelae to a fracture, conducted at all public and private orthopedic departments in Denmark, this includes 36 sites corresponding to a total of 39 departments.

DETAILED DESCRIPTION:
The outcome measures will be extracted from the following national databases: The Civil Registration System (CRS), The Danish Hip Arthroplasty Register (DHR), The Danish National Patient Registry (DNRP), The Hospital Acquired Infections Database (HAIBA), The Danish National Prescription Database (NPR), Statistics Denmark and Danish Agency for Labour Market and Recruitment registry (STAR).

Details regarding the Arms and Interventions:

The preoperative dose of antibiotic must be administered prior to surgical incision and in cases of delay with regards to planned surgical incision:

Dicloxacillin/Cloxacillin: If the preoperative antibiotic dose is administered >60 minutes prior to surgical incision, the initial dose must be repeated.

Cefuroxime: If the preoperative antibiotic dose is administered >90 minutes prior to surgical incision, the initial dose must be repeated.

Treatment A, Single-dose practice:

For patients ≥ 120 kg:

One preoperative single dose of either Dicloxacillin/Cloxacillin 3g OR Cefuroxime 3g administered intravenously prior to surgical incision.

In cases of cephalosporin allergy or general beta lactam allergy one preoperative single dose of Clindamycin 900mg administered intravenously, prior to surgical incision, regardless of weight.

Treatment B, Multiple-dose practice:

For patients ≥ 120 kg:

One preoperative single dose of either Dicloxacillin/Cloxacillin 3g OR Cefuroxime 3g administered intravenously prior to surgical incision, followed by 3 postoperative doses of Dicloxacillin/Cloxacillin 2g x 3 OR cefuroxime 1.5g x 3, administered within 24 hours after the preoperative dose, corresponding to 6, 12 and 18 hours postoperatively.

After the first postoperative dose, the remaining doses may be administered perorally for pragmatic reasons.

Dicloxacillin p.o. 1g, 12 and 18 hours postoperatively. OR Amoxicillin and clavulanic acid p.o. 875mg/125*mg, 12 and 18 hours postoperatively.

*If the center or region does not have access to amoxicillin and clavulanic acid 875/125mg a dose of 1g / 125mg (this means amoxicillin 500mg + amoxicillin and clavulanic acid 500mg/125 mg) may be administered.

In cases of cephalosporin allergy or general beta lactam allergy one preoperative single dose of Clindamycin 900mg administered intravenously, prior to surgical incision, regardless of weight, followed by 2 postoperative doses corresponding to:

For patients <120kg: 300mg, 8 and 16 hours postoperatively. For patients ≥ 120kg: 600mg, 8 and 16 hours postoperatively. The same doses apply in cases of transmission to peroral antibiotics.

Implementation: The senior biostatistician is responsible for the randomization process of the centers. Each center will be allocated a code by the senior biostatistician responsible and reported to a central database. The randomization and allocation procedure will be known for the given year conditioning the given center.

Ethics and Dissemination: This trial has been approved by the Regional Ethical Committee (VEK) (21069108) and The Danish Medicines Agency (2021091723) without imposing an obligation to notify.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving a primary Total Hip Arthroplasty (THA) due to an acute- or sequelae of proximal femoral or acetabular fractures

Exclusion Criteria:

* Patients receiving a primary THA due to bone tumor or metastasis
* Patients receiving a primary THA due to osteoarthritis and all reasons according to the Danish Hip Arthroplasty Register (DHR) except conditions mentioned in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Prosthetic joint infections (PJI) | Within 90 days from index surgery
  The definition of PJI is based on revision surgery. Revision surgery is defined as a new surgical intervention the first time after the primary intervention including debridement alone or in combination with complete or partial removal or exchange of the implant.
  The definition of PJI is based on revision surgery. Revision surgery is defined as a new surgical intervention the first time after the primary intervention including debridement alone or in combination with complete or partial removal or exchange of the implant.
  1. Two or more intraoperative deep-tissue samples of phenotypically indistinguishable bacteria isolated from at least 3 deep-tissue samples
  2. One or more positive intraoperative samples from a closed fluid aspirate AND a biopsy (fluid AND tissue) of phenotypically indistinguishable bacteria isolated
  3. A PJI when an indication of deep infection is reported to The Danish Hip Arthroplasty Registry (DHR) by the surgeon upon revision surgery

SECONDARY OUTCOMES:
Number of patients with one or more Serious Adverse Events (SAEs) | Within 90 days from index surgery
  SAEs are defined according to the ICH-GCP guidelines. SAE refers to an event involving a significant risk of death or disability of the patient (or their offspring), including, but not limited to, an event that:
  * results in death
  * is life-threatening - in the investigator's opinion the patient was in immediate risk of death from the adverse event when it appeared
  * requires hospitalization or prolongs existing hospitalization
  * results in permanent or significant disability
  * is a congenital anomaly SAEs are recorded from The Danish National Patient Registry (DNPR).
Incidence of Potential PJI referred to as PJI-likely | Within 90 days from index surgery
  PJI-likely is defined as at least one of the two criteria:
  1. One single intraoperatively obtained positive culture (aspiration fluid OR tissue biopsy) regardless of microorganism
  2. One single positive culture obtained from aspiration of synovial fluid regardless of microorganism AND any antibiotic prescriptions (ATC category J01) redeemed
Length of hospital stay (LOS) | Within 90 days from index surgery
  LOS defined as number of postoperative overnight stays, including transferals to other departments and hospitals. Data on LOS is acquired from DNPR.
Incidence of Major Adverse Cardiovascular Events (MACE) | Within 90 days from index surgery
  A MACE is defined a priori to include thromboembolic complications including venous thromboembolism, myocardial infarction, atrial fibrillation and stroke based on the diagnostic ICD10 codes listed in Appendix B. VTE is defined a priori as both deep venous thromboembolisms confirmed by compression ultrasound and pulmonary embolism confirmed by spiral computed tomography (CT), ventilation-perfusion scintigraphy or pathological removal of an embolus and based on the following diagnostic ICD10 codes: I26, I80.1-I80.9, I82.1-I82.9, or T81.7B-D. Data will be extracted from DNPR.
Hospital-treated infections (excluding Surgical Site infections) | Within 90 days from index surgery
  Any Hospital-treated infection is defined as any first-time hospital admission with a primary or secondary infection diagnosis after discharge from index THA surgery. Hospital-treated infections are identified from DNPR.
  The list of infections includes chronic and more rare infections, to detect possible flare-up in any possible ongoing infections.
  The list will exclude urinary tract infections (UTI) due to a high risk of different registration praxis registration for UTI among hospitals in Denmark.
Proportion of patients with at least one dispensing for antibiotic | Within 90 days from index surgery
  Community-based antibiotic use (any community-treated infection or antibiotic use after discharge) is defined as at least one dispensing after discharge from index THA surgery within 90 days for narrow- and broad-spectrum antibiotics based on the Anatomical Therapeutic Chemical classification (ATC) codes. All antibiotics in Denmark require prescriptions from a physician. The Danish National Health Service Prescription Database has registered all reimbursed prescriptions from all community pharmacies since 2004. Medications are coded according to the following ATC codes: J01CE, J01CF, J01DB, J01DC, J01DD, J01DE, J01DH, J01DI, J01CR, J01CA, J01F. J01E, J01MA ,J01AA
Opioid use | Within 90 days from index surgery
  Prescriptions will be identified using NPR. The following ATC codes (including all subcodes) are included: N01AH (opioid anesthetics), N02A (opioids), N07BC02 (methadone), and R05DA04 (codeine). We defined opioid users as patients who redeemed two opioid prescriptions within six months prior to THA surgery. Conversely, patients who did not redeem two or more opioid prescriptions within this timeframe were classified as opioid naïve. For opioid naïve patients, opioid use post-THA is defined as the redemption of two opioid prescriptions within 90 days following surgery. We assert that two separate redeemed prescriptions confirm actual medication use. We will calculate the treatment dosage based on the number of packages and volume redeemed within 90 days post-surgery. To investigate dosages, all doses will be converted to morphine milligram equivalents using a conversion factor specific to the type of opioid.
Use of acetaminophen or non-steroidal anti-inflammatory drugs | Within 90 days from index surgery
  Patients who received at least one prescription for acetaminophen or nonsteroidal anti-inflammatory drugs (NSAIDs) following THA surgery. Prescriptions of analgesics will be identified using NPR (41). All analgesics in Denmark except 10-tablet packages of acetaminophen / ibuprofen of dose 200mg ibuprofen require prescriptions from a physician. Following ATC codes (including all subcodes) are included M01A (NSAIDs) and N02BE01 (paracetamol). Duration of treatment will be calculated based on number of packages and volume. Since there is no clear definition of acetaminophen or non-steroidal anti-inflammatory users, we define these users as patients who redeemed two prescriptions within 6 months before THA.
Any revision after THA | Within 90 days from index surgery
  Revision surgery is defined as a new surgical intervention the first time after the primary intervention including debridement alone or in combination with complete or partial removal or exchange of any implants. Rate of revision is defined as revision due to any cause within 90 days from primary THA surgery. Any revision will be recorded from DHR and DNPR.

OTHER OUTCOMES:
Incremental cost-effectiveness | Within 90 days from index surgery
  The incremental cost-effectiveness will be calculated based on the costs per patient in the two antibiotic practices. Costs related to antibiotic prophylaxis, hospital admissions and readmissions, hospital outpatient visits, visits to General practitioner and costs related to sick leave from work will be included.
  Data will be collected from:
  * The Danish National Patient Registry (DNPR)
  * The Civil Registration System (CRS)
  * The Danish Agency for Labor Market and Recruitment registry STAR
Rate of revision after THA | Within 1 year from index surgery
  Revision surgery is defined as a new surgical intervention the first time after the primary intervention including debridement alone or in combination with complete or partial removal or exchange of the implant. Revision due to any cause including PJI and aseptic loosening are included.
  Revision risk is recorded from DHR and DNPR.
Mortality rate after index surgery | Within 1 year from index surgery
  1-year mortality rate is defined by date of death due to any cause after index surgery. Data is collected from The Civil Registration System (CRS).
Incidence of Superficial incisional Surgical Site Infection | Within 90 days from index surgery
  To be defined

CONTACTS AND LOCATIONS:
Overall Officials: Armita A Abedi, MD, Principal Investigator — Copenhagen University Hospital, Bispebjerg Department of Orthopedic Surgery and Traumatology
Locations (36):
- Denmark (36):
  - Department of Orthopedic Surgery, Aabenraa and Sønderborg, Hospital of Southern Jutland, Aabenraa
  - Capio Private Hospital, Aalborg, Aalborg
  - Department of Orthopedic Surgery, Aalborg, Aalborg University Hospital, Aalborg
  - Aleris Private Hospital, Aarhus, Aarhus
  - Deaprtment of Orthopaedic Surgery, Aarhus University Hospital, Aarhus
  - Capio Private Hospital, Aarhus, Aarhus C
  - Capio Private Hospital, Gildhøj, Brøndby
  - Department of Orthopedic Surgery and Traumatology, Bispebjerg, Copenhagen University Hospital - Bispebjerg and Frederiksberg, Copenhagen NV
  - Adeas Private Hospital, Parken, Copenhagen Ø
  - Department of Orthopedic Surgery, Esbjerg, Hospital of South West Jutland, Esbjerg
  - Department of Orthopedic Surgery, Farsø, Aalborg University Hospital, Farsø
  - CPH Private Hospital, Farum
  - Department of Orthopedic Surgery, Frederikshavn, Aalborg University Hospital, Frederikshavn
  - Department of Orthopedic Surgery, Grindsted, Hospital of South West Jutland, Grindsted
  - Capio Private Hospital, Hellerup and Odense, Hellerup
  - Department of Orthopaedic Surgery, Gentofte, Copenhagen University Hospital - Herlev and Gentofte, Hellerup
  - Department of Orthopaedic Surgery, Herlev, Copenhagen University Hospital - Herlev and Gentofte, Herlev
  - Department of Orthopedic Surgery, Gødstrup Regional Hospital, Herning
  - Department of Orthopedic Surgery, Hillerød, Copenhagen University Hospital - North Zealand, Hillerød
  - Department of Orthopedic Surgery, Copenhagen University Hospital - Holbæk, Holbæk
  - Department of Orthopedic Surgery, Horsens Regional Hospital, Denmark, Horsens
  - Department of Orthopedic Surgery, Hvidovre, Copenhagen University Hospital - Amager and Hvidovre, Hvidovre
  - Acure Private Hospital, Kongens Lyngby
  - Kollund Private Hospital, Kollund, Kruså
  - Department of Orthopedic Surgery, Zealand University Hospital, Køge, Køge
  - Department of Orthopedic Surgery, Copenahegn University Hospital - Nykøbing F., Nykøbing Falster
  - Department for Planned Orthopaedic Surgery, Næstved, Copenhagen University Hospital - Næstved, Slagelse and Ringsted, Næstved
  - Department of Orthopedic Surgery and Traumatology, Odense University Hospital and Svendborg Hospital, Odense
  - Deparmtent of Orthopedic Surgery, Randers Regional Hospital, Randers
  - Aleris Private Hospital, Ringsted, Ringsted
  - Department of Surgery, Copenhagen University Hospital - Bornholm, Rønne
  - Center for Planned Surgery, Silkeborg Regional Hospital, Silkeborg
  - Aleris Private Hospital, Søborg, Søborg
  - Department of Orthopedics, Lillebaelt Hospital, Vejle, Vejle
  - Mølholm Private Hospital, Vejle, Vejle
  - Deparmtent of Orthopedic Sugery, Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
Access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), will be provided to anyone who wishes to access the data.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication, no end date.
Access Criteria: Anyone who wishes to access the data.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT05530174/SAP_000.pdf